CLINICAL TRIAL: NCT01067807
Title: Proellex Pharmacokinetics Bridging Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZP-001
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Pharmacokinetics
MeSH Terms: interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Proellex Formulation 1 (Experimental): 25 mg Proellex Gelucire and PEG (original formulation)
  Interventions: Drug: 25 mg Proellex
- 25 mg Proellex Formulation 2 (Experimental): 25 mg Proellex coated with MCC
  Interventions: Drug: 25 mg Proellex
- 25 mg Proellex Formulation 3 (Experimental): 25 mg Proellex blended with MCC
  Interventions: Drug: 25 mg Proellex
- 50 mg Proellex Formulation 3 (Experimental): 50 mg Proellex blended with MCC
  Interventions: Drug: 50 mg Proellex

INTERVENTIONS:
Drug: 25 mg Proellex — 25 mg - given as one 25 mg capsule (252 mg of Gelucire and 88 mg of PEG400, original formulation) [Original], single dose
  Other Names: CDB-4124; Telapristone acetate
  Arms: Proellex Formulation 1
Drug: 25 mg Proellex — 25 mg - given as one 25 mg capsule (coated with microcrystalline cellulose, new formulation) (coated), single dose
  Other Names: CDB-4124
  Arms: 25 mg Proellex Formulation 2
Drug: 25 mg Proellex — 25 mg - given as one 25 mg capsule (blended with microcrystalline cellulose, new formulation) [Blended], single dose
  Other Names: CDB-4124
  Arms: 25 mg Proellex Formulation 3
Drug: 50 mg Proellex — 50 mg - given as two 25 mg capsules (blended with microcrystalline cellulose, new formulation) [Blended], single dose
  Other Names: CDB-4124
  Arms: 50 mg Proellex Formulation 3

SUMMARY:
Healthy female subjects received a single dose of four different types of Proellex, the original 25 mg dose and three new formulations

DETAILED DESCRIPTION:
Healthy female subjects received a single dose of four different types of Proellex, the original 25 mg dose and three new formulations (24 and 50 mg dose). Blood was collected pre-dose, at specified intervals and 24 hours post dose. Each dose was separated by at least one week interval from the previous dose.

ELIGIBILITY:
Inclusion Criteria:

* Medically normal subjects with no significant abnormal findings at the screening physical examination as evaluated by the clinical Investigator
* Subject was willing to remain in the clinic for the screening visit; and for the treatment visits (day -1, day of treatment and day 1; approximately 36 hrs per treatment visit)

Exclusion Criteria:

* Post-menopausal women,
* Subject with documented endometriosis
* Subject with known uterine fibroids or vaginal polyps

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Proellex peak plasma concentration (Cmax) | 24 hours
Proellex time to peak plasma concentration (tmax). | 24 hours

SECONDARY OUTCOMES:
The area under the plasma concentration over time curve from zero to the last measurable Proellex plasma concentration (AUC0-24) was calculated. | 24 hours
The area under the plasma concentration over time curve from zero to infinity (AUC 0-infinity). | 24 hours
Terminal elimination half-life (t1/2). | 24 hours
Vital signs evaluated at screening, treatment days 0 and 1. Clinical laboratory values obtained at screening, treatment days 0 and 1. Adverse events assessed at treatment visits and followed until resolution. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andre van As, PhD, MD, Study Director — Repros Therapeutics Inc.
Locations (1):
- Healthcare Discoveries, Inc, San Antonio, Texas, United States